CLINICAL TRIAL: NCT03440827
Title: Development and Validation of a Specific Scale of Life'Quality for Children With Low-flow Vascular Malformations Aged 11 to 15 Years-old.
Brief Title: Development of a Specific Scale of Life'Quality for Children With Low-flow Vascular Malformations
Acronym: MVFL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0210; 2017-A01881-52 (Other: UHToulouse)
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Vascular Malformations
Keywords: low-flow vascular malformations, scale of life's quality
MeSH Terms: conditions — Vascular Malformations | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Child with slow-flow malformation (Other): Phase 1: Collect of experiences, perceptions, difficulties, needs and expectations of patients with slow-flow vascular malformation (for the age group of 11 to 15 years-old) using the focus group method.
  Phase 2 : Administration of the scale of life's quality for validation.
  Interventions: Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Focus Group — First (phase 1), collect experiences, perceptions, difficulties, needs and expectations of patients with slow-flow malformations (for the age group of 11 to 15 years-old), carried out with 3 categories of participants and then (phase 2) development and validation of the specific scale of life's quality of slow-flow vascular malformation in children aged 11 to 15 years-old.

SUMMARY:
The low-flow malformations include venous and lymphatic malformations. The malformation often affects the skin and can extend deep to the muscles and bone, as well as to deep organs. Children with low-flow vascular malformation and their family have difficulty living with their illness and have an impact on their life quality.

In this context, the aim of the study is to develope life quality test for the children between 11 to 15 years old.

DETAILED DESCRIPTION:
The low-flow vascular malformations include venous and lymphatic malformations. These malformations are made of dilated dysplastic vessels in which the circulation is lowed down, which can lead to phenomena of thrombosis, hemorrhage, with sometimes a repercussion on the general coagulation. The malformation often affects the skin and can extend deep to the muscles and bone, as well as to deep organs. It presents by swelling sometimes voluminous and often painful. Children with low-flow malformations and their families have difficulty living with their illness and have an impact on their quality of life (QOL).

These difficulties seem relative to :

* the lack of knowledge of the disease by doctors and the general public - medical difficulties directly related to the disease and its evolution: pain, deformation, biological anomaly, chronicity, lack of effective treatment
* psychological difficulties related to the visible and unesthetic appearance of the lesions
* excluding certain social activities The difficulties experienced by patients with slow-flow malformations and their family, as well as the impact on their QOL, have never been studied. Although QOL appears to be the best reflection of the severity of a chronic condition, there is no QOL questionnaire that is appropriate for the slow-flow malformations of the child or adult.

The aim of the study is to develope a specific life quality test for children between 11 to 15 years old.

These data will be used in a second time to build and validate a scale of quality of life specific slow-flow malformations of the child aged 11 to 15 years old. The study is build in 3 parts:

Focus group: collect the dimension of the lived experience and the perceptions of the children with slow-flow malformations as well as their needs and their expectations

Validation of the life quality test: the data obtained during focus group will be used to develop the scale of life quality specific to the child aged 11 to 15 years suffering to low-flow malformations. In a second time to validate the scale, this life quality test will be send to patients.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Patient with slow-flow vascular malformation, regardless of clinical form, severity (clinical and imaging diagnosis), aged 11 to 15 years-old.
* Patient with slow-flow vascular malformation, whatever its clinical form, its severity (clinical and imaging diagnosis), aged over 15 years-old.
* Parents of a patient with slow-flow vascular malformation, regardless of clinical form, severity (clinical and imaging diagnosis), aged 11 to 15 years-old inclusive
* Patient affiliated to a social security scheme
* Patient having given his consent or for the minor whose legal representative has given written informed consent.

Phase 2 :

* Patient with slow-flow vascular malformation, regardless of clinical form, severity (clinical and imaging diagnosis), 11 to 15 years-old of age included.
* Patient affiliated to a social security scheme
* Patient having given his consent or for the minor whose legal representative has given his informed consent

Exclusion criteria :

For both phases: Pregnant or lactating women or girls,

* Vulnerable persons,
* Majors subject to a legal protection measure or unable to express their consent Phase 1: Patient or parent who does not speak the French language and therefore are unable to express themselves in the focus groups.
* Patient under 11 years-old; Phase 2 : Patient who does not speak French and is therefore unable to complete quality of life questionnaires
* Patient under 11 or over 15 years-old.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Specific scale of life's quality for slow-flow vascular malformation | 12 months
  Specific scale of life's quality for slow-flow vascular malformation.
  * the preliminary version of which is created by transforming the qualitative categories resulting from the qualitative analysis of the verbatim into an exhaustive list of thematic items which will then be selected and sorted by the experts
  * and whose final version is obtained by the statistical validation analysis aimed at structural validity and unidimensionality and convergent and discriminant validity.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Mazereeuw-Hautier, MD, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - UHBordeaux, Bordeaux
  - UHChambray, Chambray-lès-Tours
  - UHNantes, Nantes

IPD SHARING:
Plan to Share IPD: No